CLINICAL TRIAL: NCT01402375
Title: Comparing the Efficacy of Oral Opioids for Outpatient Acute Pain Management After ED Discharge
Brief Title: Comparing the Efficacy of Oral Opioids for Outpatient Acute Pain Management After ED Discharge Discharge
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, PI, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-02-066
Record Dates: First submitted 2011-07-24; First posted 2011-07-26 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Analgesia After ED Discharge for Extremity Injuries
Keywords: Pain Management; Emergency Medicine; Extremity Injuries
MeSH Terms: conditions — Agnosia | interventions — Hydrocodone; acetaminophen, hydrocodone drug combination; Acetaminophen; Codeine; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Hydrocodone (first trial) (Experimental): Hydrocodone 5mg / Acetaminophen 500mg. Patients instructed to take 1 dose every 4 hrs as needed for pain.
  Interventions: Drug: Hydrocodone (first trial)
- Codeine (first trial) (Active Comparator): Codeine 30mg / Acetaminophen 300mg. Patients instructed to take 1 dose every 4 hrs as needed for pain.
  Interventions: Drug: Codeine (first trial)
- Oxycodone (for second trial) (Experimental): Oxycodone 5mg / Acetaminophen 325mg. Patients instructed to take 1 dose every 4 hrs as needed for pain.
  Interventions: Drug: Oxycodone (for second trial)
- Codeine (for second trial) (Active Comparator): Codeine 30mg / Acetaminophen 300mg. Patients instructed to take 1 dose every 4 hrs as needed for pain.
  Interventions: Drug: Codeine (for second trial)
- Oxycodone (third trial) (Experimental): Oxycodone 5mg / Acetaminophen 325 mg. Patients instructed to take 1 dose every 4 hours as needed for pain.
  Interventions: Drug: Oxycodone (third trial)
- Hydrocodone (third trial) (Active Comparator): Hydrocodone 5mg / Acetaminophen 325 mg. Patients instructed to take 1 dose every 4 hours as needed for pain.
  Interventions: Drug: Hydrocodone (third trial)

INTERVENTIONS:
Drug: Hydrocodone (first trial) — Patients will take 1 dose of Hydrocodone 5mg / Acetaminophen 500mg every 4 hours as needed for pain
  Other Names: Vicodin (Hydrocodone 5mg / Acetaminophen 500mg)
  Arms: Hydrocodone (first trial)
Drug: Codeine (first trial) — Patients will take 1 dose of Codeine 30 mg / Acetaminophen 300 mg every 4 hours as needed for pain
  Other Names: Tylenol # 3 (Codeine 30 mg/Acetaminophen 300 mg)
  Arms: Codeine (first trial)
Drug: Oxycodone (for second trial) — Patients will take 1 dose of Oxycodone 5 mg / Acetaminophen 325 mg every 4 hours as needed for pain
  Other Names: Percocet (Oxycodone 5mg/Acetaminophen 325 mg)
  Arms: Oxycodone (for second trial)
Drug: Codeine (for second trial) — Patients will take 1 dose of Codeine 30 mg / Acetaminophen 300 mg every 4 hours as needed for pain
  Other Names: Tylenol # 3 (Codeine 30 mg/Acetaminophen 300 mg)
  Arms: Codeine (for second trial)
Drug: Oxycodone (third trial) — Patients will take 1 dose of Oxycodone 5mg / Acetaminophen 325 mg every 4 hours as needed for pain
  Other Names: Oxycodone 5mg / Acetaminophen 325 mg
  Arms: Oxycodone (third trial)
Drug: Hydrocodone (third trial) — Patients will take 1 dose of Hydrocodone 5 mg / Acetaminophen 325 mg every 4 hours as needed for pain.
  Other Names: Hydrocodone 5mg / Acetaminophen 325 mg
  Arms: Hydrocodone (third trial)

SUMMARY:
There will be 3 randomized, double-blinded clinical trials to help determine which of commonly prescribed oral opioid combination is most effective in managing acute extremity pain after discharge from the adult emergency department. The first trial compares hydrocodone 5mg / acetaminophen 500mg to codeine 30mg/acetaminophen 300mg. The second trial compares oxycodone 5mg/acetaminophen 325mg to codeine 30mg/acetaminophen 300mg. The third trial compares oxycodone 5mg/acetaminophen 325 mg to hydrocodone 5mg/acetaminophen 325 mg.

DETAILED DESCRIPTION:
Eligible patients are those between the ages of 21 and 64 who present to the Emergency Department (ED) with a complaint of acute extremity pain of less than seven days duration in one or more extremities and for whom the clinician plans to discharge on an oral opioid for pain management. Patients will be excluded if they have ever taken methadone; have a chronic condition requiring frequent pain management such as sickle cell disease, fibromyalgia, or any neuropathy; report a history of an adverse reaction to any of the study medications; if they have taken prescribed opioids in the past 24 hours or if they report having ever taken recreational narcotics; if they have a medical condition that might affect their metabolism of opioid analgesics or acetaminophen; or if they take any medicine that might interact with one of the study medications. Patients will be referred by the attending physician or clinician and consent as well as the initial and follow-up data collections will be obtained by our team of trained bilingual (Spanish and English) salaried research associates who staff the ED 24 hours a day and 7 days a week.

In the first study, patients will be randomized to one of two experimental groups: hydrocodone 5mg / acetaminophen 500mg or codeine 30mg / acetaminophen 300mg. Randomization will be performed in blocks of 10 and determined by a sequence generated at http://www.randomization.com. The pharmacist working in an area inaccessible to ED staff will ensure proper blinding of the study by masking the medication and inserting it into unmarked gel capsules and filling any void with small amounts of lactose. A three-day supply (18 doses) of the blinded medications will be dispensed by the ED staff to the patient in the order determined by randomization accompanied by instructions to use one tablet of the medication every 4 hours as needed for pain and to avoid use of any other analgesics.

Using a power of 80%, a significance criterion of 0.5, and an estimated delta of 1.3 NRS units, a sample size of 85 patients per group. In order to account for those that do not end up taking the medicine, it is estimated that 120 patients per group will have to be enrolled.

Data will be collected on a standardized data collection instrument, entered by a trained data clerk, and reviewed and audited for accuracy and completeness. The investigators will calculate descriptive statistics for all variables: frequencies, means and standard deviations, medians and IQR, and proportions. Chi-square tests will be used to test differences between dichotomous variables, t-tests will be used to test mean differences. Multivariate models will be used if there are background variables that are unevenly distributed between the two groups. Variables associated with group membership with probability of 0.20 or less will be included in OLS multivariate regression or logistic regression models in order to test the role of group membership while accounting for chance baseline disparities. Interaction terms will be tested and dropped from the models if they were not statically significant at the 0.05 level. SPSS version 17 (Chicago, IL.) will be used to conduct all data analyses.

The second trial will be identical to the first trial with the exception of one of the study drugs, which will be oxycodone 5mg / acetaminophen 325 mg which will be compared to codeine 30mg / acetaminophen 300mg.

The third trial will be identical to the first and second trials with the exception of study drugs. This study will use oxycodone 5 mg/acetaminophen 325mg and hydrocodone 5mg/acetaminophen 325mg.

ELIGIBILITY:
Inclusion Criteria:

* patient has complaint of acute extremity pain (less than 7 days duration)
* clinician plans to discharge on oral pain medication

Exclusion Criteria:

* patients on methadone
* chronic pain condition such as sickle cell anemia or fibromyalgia
* history of adverse reaction to one of the study medications
* taken prescribed opioids in the past 24 hrs
* have a medical condition that might alter the metabolism of one of the study medications (i.e. hepatitis, renal insufficiency, thyroid disease, Adrenal disease)
* Take a medication that might interact with one of the study medications

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Chang, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
Started | 120 | 120 | 120 | 120 | 120 | 120
Completed | 120 | 120 | 120 | 120 | 120 | 120
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients excluded from data analysis:
  First trial - patients did not take study medication Second trial - 7 patients unable to be reached for follow up, 18 did not take study medication Third trial - 5 patients unable to be reached for follow up, 15 did not take study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial) | Total
Number analyzed (Participants) | 88 | 93 | 111 | 104 | 107 | 113 | 616
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (12) | 37 (11) | 39 (12) | 38 (11) | 39 (12) | 38 (13) | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 48 | 62 | 58 | 60 | 48 | 314
  Male | 50 | 45 | 49 | 46 | 47 | 65 | 302
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 56 | 69 | 66 | 71 | 67 | 73 | 402
  African American | 27 | 18 | 35 | 27 | 32 | 28 | 167
  Other | 5 | 6 | 10 | 6 | 8 | 12 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 93 | 111 | 104 | 107 | 113 | 616
NRS pain intensity score on ED arrival [Median (Inter-Quartile Range); unit: units on a scale] — Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable")
  units on a scale | 9 [8 to 10] | 9 [8 to 10] | 10 [8 to 10] | 10 [8 to 10] | 10 [8 to 10] | 10 [8 to 10] | 10 [8 to 10]
NRS pain intensity score on discharge [Median (Inter-Quartile Range); unit: units on a scale] — Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable").
  The study involved patients taking study medications AFTER emergency department discharge, and the primary outcome also involved NRS pain scores 24 hours AFTER ED discharge. Thus, any data collected while in the ED is considered baseline.
  units on a scale | 7 [5 to 8] | 7 [5 to 8] | 7 [6 to 9] | 7 [5 to 9] | 8 [6 to 9] | 8 [6 to 9] | 7 [5 to 9]
Diagnosis [Count of Participants; unit: Participants]
  Sprain/strain | 40 | 54 | 59 | 49 | 39 | 42 | 283
  Extremity Fracture | 20 | 17 | 33 | 37 | 63 | 58 | 228
  Other | 28 | 22 | 19 | 18 | 5 | 13 | 105
Took analgesic prior to presentation [Count of Participants; unit: Participants]
  No | 63 | 63 | 72 | 70 | 76 | 74 | 418
  Yes | 24 | 27 | 37 | 33 | 29 | 36 | 186
  Unknown | 1 | 3 | 2 | 1 | 2 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Difference in Pain Intensity Score Before and After Last Dose.
Description: Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable"). The difference in pain score is calculated by subtracting the average score 2 hours after pain medication is taken from the average pain score immediately before the pain medication is taken.
Time Frame: 2 hrs
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
Number analyzed (Participants) | 88 | 93 | 111 | 104 | 107 | 113
units on a scale
  before most recent dose | 7.6 (1.7) | 7.6 (1.8) | 7.9 (1.5) | 7.9 (1.7) | 7.8 (1.5) | 7.6 (1.6)
  2 hours after most recent dose | 3.6 (2.8) | 4.1 (2.9) | 3.4 (2.5) | 3.6 (4.2) | 3.3 (2.7) | 3.6 (2.6)
  change in NRS before to after most recent dose | 3.9 (2.5) | 3.5 (2.6) | 4.5 (2.4) | 4.2 (2.4) | 4.4 (2.5) | 4.0 (2.5)

2. Secondary Outcome: Overall Satisfaction With the Pain Medicine
Description: Overall satisfaction with the oral opioid pain medication at 24 hours after discharge using a Likert scale. Patients will be asked to describe their overall experience as being very satisfied, satisfied, unsatisfied or very unsatisfied with the study medication.
Time Frame: 24 hrs
Population: Any number analyzed that does not equal the overall number of participants is due to missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
Number analyzed (Participants) | 88 | 93 | 111 | 104 | 107 | 113
Participants
  Number of participants satisfied with analgesic: number analyzed (Participants) | 87 | 93 | 111 | 104 | 107 | 113
  Number of participants satisfied with analgesic | 72 | 66 | 99 | 91 | 93 | 97
  participants would want the same analgesic again: number analyzed (Participants) | 85 | 93 | 111 | 104 | 107 | 113
  participants would want the same analgesic again | 59 | 66 | 91 | 85 | 86 | 90

3. Post Hoc Outcome: 50% or Greater Decrease in Numerical Rating Scale (NRS) Pain Score
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
Number analyzed (Participants) | 88 | 93 | 111 | 104 | 107 | 113
Participants | 50 | 45 | 73 | 64 | 68 | 66

4. Post Hoc Outcome: Time to Follow up
Description: Median time to contact patients for data collection, measured from discharge to time contacted
Time Frame: up to 48 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
Number analyzed (Participants) | 88 | 93 | 111 | 104 | 107 | 113
hours | 27 [24 to 42] | 25 [24 to 36] | 26 [24 to 37] | 28 [25 to 36] | 27 [25 to 42] | 28 [25 to 41]

ADVERSE EVENTS:
Time Frame: follow up period, 24-48 hours
Description: In adverse events, any change in total participants at risk from overall number reflects missing data
Arm/Group | Hydrocodone (First Trial) | Codeine (First Trial) | Oxycodone (for Second Trial) | Codeine (for Second Trial) | Oxycodone (Third Trial) | Hydrocodone (Third Trial)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/93 | 0/111 | 0/104 | 0/107 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/93 | 0/111 | 0/104 | 0/107 | 0/113
Other Adverse Events (participants affected / at risk) | 54/88 | 51/93 | 68/111 | 61/104 | 74/106 | 51/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Hydrocodone (First Trial) (N=88) | Codeine (First Trial) (N=93) | Oxycodone (for Second Trial) (N=111) | Codeine (for Second Trial) (N=104) | Oxycodone (Third Trial) (N=106) | Hydrocodone (Third Trial) (N=112)
Nausea (Gastrointestinal disorders) | 9/87 | 9/92 | 13 | 12 | 18/105 | 8
Vomiting (Gastrointestinal disorders) | 2/87 | 1/92 | 4 | 2 | 5/105 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2/110
Diarrhea (Gastrointestinal disorders) | 0/87 | 5 | 1 | 3 | 3 | 2/110
Pruritus (Skin and subcutaneous tissue disorders) | 3/87 | 3 | 6 | 4 | 3 | 4/110
Rash (Skin and subcutaneous tissue disorders) | 1/87 | 0/92 | 2 | 3 | 2 | 2/111
Dizziness (Nervous system disorders) | 12/87 | 5 | 11 | 13 | 18 | 8/111
Drowsiness (Nervous system disorders) | 25 | 27 | 30 | 23 | 24/105 | 23
Confusion (Nervous system disorders) | 2/86 | 1 | 1 | 1 | 1/104 | 1/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes